CLINICAL TRIAL: NCT04663542
Title: A Prospective Randomized Controlled Clinical Trial on the Comparison of the Treatment Outcomes of Different Immobilization Times After the Repair of Achilles Tendon Rupture
Brief Title: The Efficacy of Different Immobilization Times After Achilles Tendon Rupture Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUTH LY ATR; 81702127 (Other Grant/Funding Number: National Natural Science Foundation of China); 2018YFF0301100 (Other Grant/Funding Number: Science and Technology fund of Winter Olympics)
Record Dates: First submitted 2020-09-16; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-09

CONDITIONS: Achilles Tendon Rupture
Keywords: immobilization duration; open surgery; early rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0-week immobilization (Experimental): 0-week brace immobilization after the surgery will be conducted.
  Interventions: Procedure: immobilization duration
- 2-week immobilization (Experimental): 2-week brace immobilization after the surgery will be conducted.
  Interventions: Procedure: immobilization duration
- 4-week immobilization (Other): 4-week brace immobilization after the surgery will be conducted.
  Interventions: Procedure: immobilization duration
- 6-week immobilization (Other): 6-week brace immobilization after the surgery will be conducted.
  Interventions: Procedure: immobilization duration

INTERVENTIONS:
Procedure: immobilization duration — brace immobilization duration after open surgery for Achilles tendon rupture

SUMMARY:
This study is a prospective randomized controlled clinical study. After the Achilles tendon rupture repaired by our suture technique, patients were randomly divided into 4 groups, and the brace fixation time was 0, 2, 4 and 6 weeks, respectively, to study the difference in efficacy between the groups.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical study is designed to compare the treatment outcomes of different immobilization times by dividing the patients into four groups-A, B, C, and D-based on the amount of immobilization time (0, 2, 4, and 6 weeks, respectively) that include a similar rehabilitation protocol. The inclusion criteria are patients with an acute closed single-legged complete Achilles tendon rupture, and an age of 18 to 60 years. The exclusion criteria are patients with prior Achilles tendon rupture or other situations that affect their lower limb functions or tendon healing (e.g., autoimmune disease, diabetes mellitus, systemic corticosteroid treatment). Other exclusion criteria are an inability to complete our suture technique (e.g., the distance from the rupture site to the Achilles tendon insertion is less than 3.5 cm), or those without rehabilitation or follow-up outcomes. All patients will be treated surgically with the same suture technique and undergo a similar rehabilitation protocol after the brace is removed.

ELIGIBILITY:
Inclusion Criteria:

* acute closed single-legged complete Achilles tendon rupture
* age of 18 to 60 years.

Exclusion Criteria:

* patients with prior Achilles tendon rupture or other situations that affected their lower limb functions or tendon healing (e.g., autoimmune disease, diabetes mellitus, systemic corticosteroid treatment).
* an inability to complete our suture technique (e.g., the distance from the rupture site to the Achilles tendon insertion was less than 3.5 cm)
* those without rehabilitation or follow-up outcomes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
the time of return to light sports activity | from operation to 1-year follow-up after the surgery
  when the patients are able to do jogging or rapid walk after the surgery, the time will be recorded.

SECONDARY OUTCOMES:
range of motion (ROM) recovery time | from operation to 1-year follow-up after the surgery
  the recovery time will be recorded when the ROM is similar to that of the uninjured side.
recovery time of the single-legged heel rise height (SHRH) | from operation to 1-year follow-up after the surgery
  The heel rise height is measured as the distance from the ground to the heel when the patient lift the heel while keeping the knee straight. The recovery time is noted when the SHRH is similar to that of the opposite leg.

OTHER OUTCOMES:
visual analogue scale (VAS) | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  VAS pain score is from 0 to 10, the higher score demonstrate the more severe pain.
American Orthopaedic Foot and Ankle Society (AOFAS) hindfoot score | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  The AOFAS score ranges from 0 to 100, with a healthy hindfoot receiving 100 points.
the Achilles tendon Total Rupture Score (ATRS) | 2, 4, 6, 8, 10, 12, 14, 16, 24, and 48 weeks after the surgery
  The ATRS includes 10 items; each item has a score ranging between 0 and 10 on a Likert scale, with 100 indicating no major limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao Y, Li X, Cui Z, Lv Y, Si G. Open surgery and minimally invasive repair of acute Achilles tendon rupture: stratified outcomes based on immobilization duration in a prospective cohort study. J Orthop Surg Res. 2025 Jul 12;20(1):647. doi: 10.1186/s13018-025-06019-0. PMID 40652259
- [Derived] Cao Y, Gao S, Cui Z, Fu Y, Bai L, Si G, Fan J, Lv Y, Zhou F. Comparison of different immobilisation durations following open surgery for acute achilles tendon rupture: a prospective cohort study. J Orthop Surg Res. 2024 Aug 21;19(1):497. doi: 10.1186/s13018-024-04970-y. PMID 39169350